Comparison of Prosthetic Feet for People With Syme's Amputation  $NCT04086641 \\ 06/02/2019$ 

## Data analysis plan

Variables that characterize the study sample. Summary statistics (i.e., means, standard deviations) will be calculated for all demographic and clinical characteristics. A paired t-test ( $\alpha$ =.05) will be used to assess whether SCS statistically differs between foot conditions to examine prosthetic comfort equivalence.

Biomechanical and self-reported health outcome variables. Biomechanical data will be assessed for quality using Qualisys Track Manager to identify markers, interpolate gaps, and truncate trials to data collected in the capture volume. Visual 3D software (C-Motion, Inc., Rockville, MD) will be used to filter data, build models, label gait events, and compute outcomes. Self-reported data will be scored according to developer instructions. All data will be assessed for adherence to statistical assumptions. If sufficiently normal, paired t-tests will be used to assess statistical difference between all biomechanical and health outcome variables ( $\alpha$  =.05). Adjustments for multiple comparisons will not be applied due to the pilot nature of the study. Prosthetic foot preference will be reported as percentages; participant qualitative comments will be compiled and reviewed to inform study findings and future research directions.

## Note:

Due to the advent of COVID-19, the goal number of participants (10) was not achieved. While five (5) participants were recruited, data was only collected for two (2) prior to cessation of human subjects research. As a result, inferential statistical analysis was not possible, and summary statistics (i.e., means, standard deviations) were used to compare prosthetic foot conditions for both participants.